CLINICAL TRIAL: NCT04659733
Title: Phase I Clinical Trial of Anlotinib in Progressive, Recurrent, and Refractory Sarcoma in Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yizhuo Zhang (Other)
Responsible Party: Sponsor-Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: anlotinib
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib hydrochloride (Experimental)
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib are divided into 3 dosage levels, including 8mg, 10mg, 12mg; Oral administration of anlotinib was given, qd, D1-D14; taken on an empty stomach, Every 3 weeks is a cycle, a total of 2 cycles; Starting from the first level of anlotinib, the dose will be ramped up in sequence.

SUMMARY:
The purpose is to observe and evaluate the safety and effectiveness of anlotinib in children with progressive, recurrent, and refractory sarcoma. Pharmacokinetics was also detected.

DETAILED DESCRIPTION:
Patients were enrolled according to the standard design of the Phase I study. Anlotinib are divided into 3 dosage levels, including 8mg, 10mg, 12mg; Oral administration of anlotinib was given, qd, D1-D14; taken on an empty stomach, Every 3 weeks is a cycle, a total of 2 cycles; Starting from the first level of anlotinib, the dose will be ramped up in sequence.

ELIGIBILITY:
Inclusion Criteria:

1.5years ≤ age ≤18 years old, regardless of gender;

2.ECOG performance status (PS) score: 0～1;

3.The expected survival time is more than 12 weeks;

4.Children with sarcoma confirmed by histopathology;

5.Patients who have progressed, recurrent or refractory disease after first-line treatment (failure to obtain complete or partial remission after recent treatment);

6.With measurable lesions (according to the RECIST 1.1 standard, the CT scan of tumor lesions has a long diameter ≥10mm, and the CT scan of lymph node lesions has a short diameter ≥15mm. The measurable lesions have not been treated with radiotherapy or cryotherapy);

7.The patients must recover from the acute toxic effects of all previous anticancer chemotherapy fully;

8.Myelosuppressive chemotherapy: at least 21 days after the last myelosuppressive chemotherapy (If nitrosourea was used in the early stage, the interval time is 42 days);

9.Experimental drugs or anti-cancer therapies other than chemotherapy: It is not allowed to use other experimental drugs within 28 days before the planned start of use, and it is necessary to fully recover from the clinically significant toxicity of the therapy;

10.Hematopoietic growth factors: at least 14 days after the last administration of long-acting growth factors or 3 days after the last administration of short-acting growth factors;

11.Immunotherapy: At least 42 days after completing any type of immunotherapy (except steroids), such as immune checkpoint inhibitors and tumor vaccines;

12.X-ray therapy (XRT): at least 14 days after local palliative XRT (small-scale mouth); if it is another substantial bone marrow (BM) irradiation, including pre-radio-iodinated metaiodobenformin (131I-MIBG) treatment, the interval time must end at least 42 days;

13.Stem cell infusion without total body irradiation (TBI): there is no evidence of active graft-versus-host disease, at least 56 days after transplantation or stem cell infusion;

14.Laboratory inspections during the screening period should meet the following conditions: The absolute value of neutrophils (ANC) ≥1.5×109/L (if the bone marrow is invaded, then ANC≥1.0×109/L) Platelet (PLT) ≥75×109/L (if bone marrow invades, then PLT ≥50×109/L) Bilirubin ≤1.5 times ULN Creatinine ≤ 1.5 times ULN (calculated according to the standard Cockcroft-Gault formula) ALT/AST≤3 times ULN (if there is liver metastasis, it can be relaxed to 5 times ULN)

15. During the study period, patients should be able to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits;

16. Parents/guardians of a child or young patients have the ability to understand, agree, and sign the research informed consent form (ICF) and applicable child consent form before initiating any program related procedures; Subjects can express consent (where applicable) with the consent of the parent/guardian.

Exclusion Criteria:

Patients with any of the following items will not be enrolled in this study:

1. Symptomatic brain metastases (patients with brain metastases who have completed treatment 21 days before enrollment and have stable symptoms can be enrolled, but they need to be evaluated by cranial MRI, CT, or venography to confirm that they have no symptoms of cerebral hemorrhage);
2. Imaging (CT or MRI) shows that the tumor focus is ≤ 5 mm from large blood vessels, or there is a tumor that invades local large blood vessels;
3. Patients with hypertension who are using two or more antihypertensive drugs in combination therapy;
4. Patients who suffer from the following cardiovascular diseases: Myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (including QTc interval ≥450 ms for males and ≥470 ms for females); according to NYHA standards, grade III to IV cardiac insufficiency, or the heart color Doppler ultrasound examination showed that the left ventricular ejection fraction (LVEF) <50%;
5. Patients with a history of interstitial pulmonary disease or who also suffer from the interstitial pulmonary disease;
6. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), have a bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
7. The daily volume of hemoptysis reached two teaspoons or more before enrollment;
8. Patients who have had clinically significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic hemorrhoids, hemorrhagic gastric ulcer, fecal occult blood++ and above at baseline, or vascular
9. Arterial/venous thrombosis events that occurred in the 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
10. Known existing hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, blood coagulation dysfunction, thrombocytopenia, hypersplenism, etc.);
11. Long-term unhealed wounds or fractures (pathological fractures caused by tumors are not counted);
12. Patients who received major surgery or suffered severe traumatic injury, fracture, or ulcer within 4 weeks of enrollment;
13. some factors significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
14. Abdominal fistula, gastrointestinal perforation, or abdominal abscess occurred within 6 months before enrollment;
15. Urine routine test showed urine protein ≥ ++, and confirmed 24-hour urine protein ≥ 1.0 g; Notes: Asymptomatic serous effusions can be included in the group, and symptomatic serous effusions have been actively treated symptomatically (anti-cancer drugs cannot be used for the treatment of serious effusions), and patients who are judged by the investigator can be included in the group，allow to join the group.
16. Active infections require antimicrobial treatment (for example, antibacterial drugs and antiviral drugs are required, excluding chronic hepatitis B anti-hepatitis B treatment, antifungal drug treatment);
17. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
18. Participated in other anti-tumor drug clinical trials within 4 weeks before joining the group;
19. Previously or concurrently suffering from other uncured malignant tumors, except for cured skin basal cell carcinoma, cervical carcinoma in situ, and superficial bladder cancer;
20. Within 7 days before the first administration, patients used drugs or foods known to be potent inhibitors of CYP3A4, including but not limited to: atazanavir, clarithromycin, indinavir, itraconazole, ketocon Azole, nefazodone, nelfinafil, ritonavir, saquinavir, telithromycin, acetoeandomycin, voriconazole, etc.;
21. Within 12 days before the first administration, use drugs known to be strong inducers of CYP3A4, including but not limited to: carbamazepine, phenobarbital, phenytoin, rifabutin, and rifapar;
22. Pregnant or breast-feeding women; fertility patients who are unwilling or unable to take effective contraceptive measures;
23. The investigator judges other situations that may affect the conduct of clinical research and the judgment of research results.
24. When the virological test during the screening period shows that any of the following is met:

HBsAg is positive and HBV DNA exceeds the upper limit of normal Anti-HCV positive and HCV RNA positive HIV positive

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
MTD of antinib | Time Frame: From observation up to 28 days
  Maximum tolerated dose of antinib

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter

REFERENCES:
- [Derived] Lu S, Que Y, Liu D, Sun F, Yao X, Deng L, Zhan J, Huang J, Cai R, Wang X, Zhu S, Zhen Z, Zhu J, Wang J, Zhang Y. Safety and feasibility of anlotinib in children with high risk, recurrent or refractory sarcomas: an open-label, single-centre, single-arm, phase Ia/Ib trial. EClinicalMedicine. 2025 May 23;84:103258. doi: 10.1016/j.eclinm.2025.103258. eCollection 2025 Jun. PMID 40496885